CLINICAL TRIAL: NCT05865769
Title: Impact of Pulmonary Function on Vestibular System in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Mohammed Torad, Lecturer, Kafrelsheikh University
Other Study IDs: P.T/PED/2/2023/41
Record Dates: First submitted 2023-04-20; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Vestibular Disorder; Pulmonary Disease
MeSH Terms: conditions — Vestibular Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal children: Have FEV1 higher than median on their class
  Interventions: Other: Balance
- subclinical pulmonary impairment: Have FEV1 lower than median on their class
  Interventions: Other: Balance

INTERVENTIONS:
Other: Balance — measuring pulmonary and vestibular functions in all subjects

SUMMARY:
The vestibular system and the pulmonary system are two critical components of the human body that are involved in maintaining balance, coordination, and the exchange of oxygen and carbon dioxide This study aim to investigate the impact of pulmonary function on the vestibular system in children.

Children aged 4 to 10 years will be recruited from Future Academy School in March 2023. Pulmonary function will be measured using digital spirometry, and balance will be evaluated using the Mini-SITCIB test, which tested vision, proprioception, and the vestibular system using mobile sensors fixed near the center of gravity. Features from the sensor data will be extracted using Python 3.10 code, and the SPSS program will used to compare these features between the two groups.

DETAILED DESCRIPTION:
The procedures of the current study will be explained to the children and their parents then parents read and sign an informed consent form.

Spirometry (spirOx plus, MEDITECH, China) will be used in the current study; Hand-held lung function test equipment uses infrared signal acquisition methods to measure the forced vital capacity-related items. It has a compact design, is lightweight and is convenient to carry and use; also, it uses low power consumption and can store up to 200 test cases. It can measure forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), peak expiratory flow (PEF) and PEF in 25%, 50%, and 75% also the device may provide percentages like FEV1/FVC, and FEP25/75. This device has proven to be valid and reliable to measure spirometry functions.

Phyphox application will be used(physical phone experiment, version 1.1.7), a free program with at least 30 functions for proceeding with physics experiments. The application is named phyphox (an acronym for physical phone experiments) and bosom on Google's Play Store and Apple's App Store in September 2016. To buttress users about the world, an accompanying website was created at http://phyphox.org, which offers itemized instructions, demonstration videos and technical information in English and German. The app itself is presently being translated into additional languages by volunteers from all around the world. The application can use the remote access option to transfer the screen to another monitor wirelessly; also, the app can measure acceleration, gyroscope, linear acceleration, and magnetometer readings. Also exporting the results is available on the wireless screen. This application is proven to be valid and reliable to measure the sensor's readings.

After obtaining the consent form, some demographic data like gender, age, weight, height and BMI were collected then each child was asked to take a deep breath and then expire for 6 sec at the spirometer.

The mobile application will be opened, and a new experiment will be created with the following criteria: sensors are acceleration, gyroscope, linear acceleration and magnetometer, the sampling rate is 800 Hz, the Experiment time is 30 sec with a 3-sec delay, then the remote access option will be enabled so that the screen appears on laptop screen wirelessly.

Abdominal support will be modified so it contains a pocket in its centre so the mobile can fit onto it. Then the mobile phone with the application opened on its screen will be fitted in the pocket in the modified belt, so when the belt is attached the mobile sensors will be very close to the centre of gravity of the participant. After wrapping the belt, participants will be asked to conduct a mini-SITCIB test. For each condition, they will be asked to stand as the condition states for 30 sec and start counting when the application starts recording the sensors data, the conditions are as follows: opened eye with the fixed surface, the closed eye with the fixed surface, opened eye with movable surface and closed eye with the movable surface. Finally, the data will be extracted and stored anonymously on the hard drive as CSV files. The condition test is over when (a) the participant opens his/her eyes in an eyes-closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall.

ELIGIBILITY:
Inclusion Criteria:

* Children will be recruited from Future Academy School. Children will be included in the current study if their age is between 4 and 10 years old, also all children are free of asthma and other respiratory diseases.

Exclusion Criteria:

* They were excluded if they had surgery or previous trauma over the chest.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children were recruited from Future Academy School. Children were included in the current study if their age is between 4 and 10 years old, also all children are free of asthma and other respiratory diseases. They were excluded if they had surgery or previous trauma over the chest. 62 children were recruited at the start of the current study; 5 children are older than the proposed sample while the parents of the other 5 refused to enter the study then the sample was classified according to FEV1 into 2 equal number classes (Low and high FEV1) according to median also 4 records were excluded as they are so extreme then the Mini-SITCIB test was used to measure balance in 4 conditions to test vision, proprioception and vestibular systems.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Root Mean Square (RMS) swaying of COG in X,Y,Z | 2 weeks
  mm
Frequency of swaying in X,Y,Z | 2 weeks
  Hz

IPD SHARING:
Plan to Share IPD: Undecided
upon request